CLINICAL TRIAL: NCT02674672
Title: A Safety and Efficacy Study for Implantation and Retrieval Procedures Using the VENATECH® Retrieval Filter System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.Braun Médical - CoE Chasseneuil (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-1419
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2016-02

CONDITIONS: Pulmonary Thrombo-embolism
Keywords: VenaTech® Retrievable Vena Cava Filter; safety; efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VenaTech Retrievable arm (Experimental): VenaTech Retrievable arm
  Interventions: Device: VenaTech® (VenaTech Retrievable Filter)

INTERVENTIONS:
Device: VenaTech® (VenaTech Retrievable Filter)

SUMMARY:
To establish the clinical safety and efficacy of the VenaTech® Retrievable Vena Cava Filter

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary thrombo-embolism with contraindication to anticoagulation.
* Failure of anticoagulant therapy in thrombo-embolic diseases.
* Prevention of pulmonary embolism in patients with a recent history ( <3 months) of DVT/ PE who need to undergo urgent surgery at high risk of DVT/PE with temporary contra-indication to the use of therapeutic doses of anticoagulants.
* Emergency treatment following massive pulmonary embolism where anticipated benefits of conventional therapy are reduced and
* Chronic, recurrent pulmonary embolism where anticoagulant therapy has failed or is contraindicated

Exclusion Criteria:

* The filter should not be implanted in patients with :

  * A vena cava which has a diameter < 14 mm or > 28 mm (due to the risk of device migration)
  * Risk of septic embolism
  * Known allergy to the materials contained in the kit, allergy to contrast media.
  * Severely disabled patients whose life-expectancy, up to 6 months, appears limited according to the investigator's opinion.

In addition, exclusion criteria are also extended to :

* Patients who cannot be regularly followed up by the participating center
* Subject who already has an implanted vena cava filter
* Subject who has a duplicated IVC
* Subject who has a contrast allergy to both iodinated contrast and non-iodinated contrast material
* Subject unable to understand information about participation in the study due to a language barrier, intellectual deficiency, psychiatric problems…
* Subject who has a renal failure (creatinemia clearance < 30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety and the efficacy of filter implantation and retrieval by the study of technical success rate of filter placement, and filter removal (when filter removal procedure is schedule) within 12 weeks of implantation | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital européen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dean C, Kim YI, Sanchez O, Martelli N, Sapoval M, Pellerin O. Safety and efficacy of the VenaTech Retrievable inferior vena cava filter: a first-in-man single-center prospective study. CVIR Endovasc. 2022 Oct 4;5(1):50. doi: 10.1186/s42155-022-00325-y. PMID 36194306